CLINICAL TRIAL: NCT06902376
Title: NEO-COMBAT XL: Neoadjuvant and Maintenance XL092 and Cemiplimab in BRAF V600E-wildtype Anaplastic Thyroid Cancer: a Phase 1B Study
Brief Title: XL092 and Cemiplimab in BRAF WT Thyroid Cancer
Acronym: NEO-COMBATXL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Regeneron Pharmaceuticals (Industry); Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2255
Record Dates: First submitted 2025-03-18; First posted 2025-03-30 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Anaplastic Thyroid Cancer; Thyroid Cancer; BRAF Mutation-Related Tumors
Keywords: neoadjuvant chemotherapy; neoadjuvant immunotherapy; standard of care; BRAF V600E-WT ATC; XL092; cemiplimab; receptor tyrosine kinase inhibitor
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic; Thyroid Neoplasms | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- neoadjuvant XL092 and cemiplimab (Experimental): Subjects with BRAFV600E wild type (WT) anaplastic thyroid cancer (ATC) who are scheduled to undergo surgical resection as part of their standard of care will receive neoadjuvant XL092 and cemiplimab. Adjuvant therapy may be indicated based on surgical pathology.
  Interventions: Biological: Cemiplimab; Drug: XL092

INTERVENTIONS:
Biological: Cemiplimab — Cemiplimab will be administered at a dose of 350mg intravenous over 30 minutes every 3 weeks for 3 cycles (cycle length is 21 days) at weeks 1, 4, and 7.
Drug: XL092 — XL092 will be administered at a dose of 60mg PO daily for 8 weeks (weeks 1-8)

SUMMARY:
This multicenter study examines the safety and feasibility of the combination of neoadjuvant XL092 and cemiplimab prior to surgical resection in participants with wild-type (WT) anaplastic thyroid cancer (ATC) that has a BRAF mutation (BRAF V600E).

DETAILED DESCRIPTION:
This study includes subjects with BRAFV600E wild type (WT) anaplastic thyroid cancer (ATC) who are scheduled to undergo surgical resection as part of their standard of care. The study hypothesizes that the combination of neoadjuvant XL092 and cemiplimab will be safe and feasible prior to surgical resection in participants with BRAF V600E-WT ATC.

Anaplastic thyroid cancer (ATC) is a highly aggressive and fatal malignancy. For patients with BRAF V600E-wildtype ATC, chemotherapy, whether as a single agent or in combination, remains the standard treatment despite its low response rates. Studies have shown that while immunotherapy (IO) and receptor tyrosine kinase inhibitor (TKI) monotherapy are safe for these patients, their efficacy as single agents is limited.

This study addresses a significant unmet need and is based on the strong synergy observed between IO and TKI in clinical studies of other cancers. It includes subjects with BRAF V600E-wildtype ATC who are scheduled for surgical resection as part of their standard care. The study hypothesizes that the combination of neoadjuvant XL092 and cemiplimab will be safe and feasible before surgical resection in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent was obtained to participate in the study and HIPAA authorization for the release of personal health information.
* Subjects are willing and able to comply with study procedures based on the judgment of the investigator.
* Age ≥ 18 years at the time of consent.
* the Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
* Pathologic findings supporting the clinical impression of anaplastic thyroid cancer. Terminology consistent or suggestive of diagnosis may include the following: anaplastic thyroid carcinoma, undifferentiated carcinoma, squamous carcinoma; carcinoma with spindled, giant cell, or epithelial features; poorly differentiated carcinoma with pleomorphism, extensive necrosis with tumor cells present.
* Subject is willing to have a fresh biopsy at least 3 days prior to neoadjuvant therapy if archival tissue is unavailable. Also willing to have a biopsy at the time of SOC surgery, if applicable.
* Must have BRAF V600E mutation-negative tumor, as determined by BRAF V600E immunohistochemistry on tumor tissue or genetic/molecular testing of the tumor.

Exclusion Criteria:

* Pregnant or breastfeeding (Note: breast milk cannot be stored for future use while the mother is being treated on the study). Females should not breastfeed while receiving study treatment and for 1 month from the last dose of XL092.
* Patients who have had prior exposure to any immune modulating agents or any type of small molecule kinase inhibitor (including investigational agents) and have documented disease progression on these agents will not be eligible.
* Ongoing or recent (within 5 years) evidence of significant autoimmune disease that required treatment with systemic immunosuppressive treatments (i.e., with use of disease modifying agents, corticosteroids (>10 mg of prednisone or equivalent) or immunosuppressive drugs) which may suggest risk of immune-mediated Adverse Events.
* Replacement therapy (e.g.: thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. The following are not exclusionary: vitiligo, childhood asthma that has resolved, type 1 diabetes, residual hypothyroidism that required only hormone replacement, or psoriasis that does not require systemic treatment.
* Subject history of documented allergic reactions or acute hypersensitivity reactions attributed to antibody treatments.
* Subject is receiving prohibited medications or treatments as listed in the protocol that cannot be discontinued/replaced by an alternative therapy within 7 days of initiating treatment.
* Participation in another clinical study with an investigational product during the last 3 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Complete gross resection | 12 weeks
  Complete gross resection (CGR) is defined as the proportion of patients who undergo successful thyroidectomy with negative (R0) or microscopically positive (R1) surgical margins.
Non-hematologic treatment related adverse events (TRAEs) | Up to 2 years
  Non-hematologic treatment related adverse events (TRAEs) with neoadjuvant and maintenance XL092 and cemiplimab will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI- CTCAE) v5.0.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 10 weeks
  Objective response rate (ORR) following neoadjuvant therapy prior to surgery as defined as a partial or complete response per Radiographic response will be measured by RECIST, 1.1 criteria. Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time to surgery | 12 weeks
  Time to surgery following completion of neoadjuvant XL092 and cemiplimab will be defined as the time from completion of neoadjuvant therapy to date of surgery. Participants who do not receive surgery due to progressive disease or non-treatment-related adverse events death will not be counted.
The rate of pathologic response | 12 weeks
  The rate of pathologic response will be defined as either a pathological complete response (pCR), which is the absence of a residual viable tumor or a major pathological response (MPR), which is < 10% residual tumor following neoadjuvant therapy and surgery.
Conversion rate from unresectable to resectable disease | 12 weeks
  Conversion rate from unresectable to resectable disease will be defined as the number of subjects with unresectable disease at the time of screening who are deemed to have resectable disease at the completion of neoadjuvant therapy.
Event free survival (EFS) | Up to 5 years
  Event free survival (EFS) will be defined as the time of first treatment to an event which may include disease progression, discontinuation of the treatment for any reason, or death from any cause, where disease progression will be determined based on RECIST 1.1 criteria. If a patient has no events, they will be censored at the last known alive date. Complete Response (CR), the disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Overall survival (OS) | Up to 5 years
  Overall survival (OS) of participants receiving neoadjuvant XL092 and cemiplimab will be defined as the time from the date of first treatment to death.

CONTACTS AND LOCATIONS:
Overall Officials: Siddharth Sheth, DO MPH, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Dana Farber/Harvard Cancer Center, Boston, Massachusetts
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials